CLINICAL TRIAL: NCT06339463
Title: Targeting Approach Behaviors in Exposures With Self-distancing to Improve Outcomes in Youth Specific Phobia
Brief Title: Self-Distancing for Specific Phobia in Youth
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding.
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Kate D. Fitzgerald, MD, Professor of Child and Adolescent Psychiatry, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAU7985
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Specific Phobias
Keywords: Self-distancing; Specific phobia
MeSH Terms: conditions — Phobia, Specific

STUDY DESIGN:
Intervention Model Description: Youth (7-12.99 years) with DSM-5 specific phobia (e.g. spider phobia) will be randomized to SD or a control condition (first-person perspective). Self-distancing or control condition will be delivered over the course of one visit. These conditions will run in parallel.
Who Masked: Outcomes Assessor
Masking Description: The rater will be blinded to which condition, self-distancing or control, child participants receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Distancing (Experimental): Youth will be randomized to a BAT with Self-Distancing Intervention. In this arm, participants will be instructed to describe the exposure task from a self-distanced perspective (e.g., "Emily is going to touch the spider").
  Interventions: Behavioral: Self-Distancing Intervention
- First-person self-talk (Active Comparator): Youth will be randomized to a BAT with a control condition. In this arm, participants will be instructed to describe the exposure task from a self-immersed perspective (e.g.,"I'm going to touch the spider")
  Interventions: Behavioral: First-person self-talk

INTERVENTIONS:
Behavioral: Self-Distancing Intervention — In the Self Distancing Intervention condition, participants will be instructed to describe the exposure task from a self-distanced perspective (e.g., "Emily is going to touch the spider").
  Arms: Self-Distancing
Behavioral: First-person self-talk — Youth will be randomized to a BAT with a control condition. In this arm, participants will be instructed to describe the exposure task from a self-immersed perspective (e.g., "I'm going to touch the spider")
  Arms: First-person self-talk

SUMMARY:
Self-Distancing is a cognitive technique that involves a shift in self-talk characterized by replacing first-person (e.g., "I") with second- or third-person pronouns (i.e., "you", one's own name) to promote an adaptive, self-reflective stance in emotionally charged situations. This trial aims to help learn how self-distancing may increase behavioral approach during exposures. To find out if self-distancing works by helping children approach fear-inducing stimuli, the study will look at behaviors and physiological responses related to approach, as well as symptom severity, before and after this cognitive technique.

The study hypothesizes that Self-Distancing will lead to greater increases in approach behaviors and a larger decrease in symptom severity compared to a control condition (first-person self-talk).

DETAILED DESCRIPTION:
Anxiety disorders impact 1 in 3 youths by the time of adolescence, and can lead to depression, substance use, school issues, and suicide risk. Specific phobia is the earliest occurring and most common anxiety disorder and increases risk for later onset of other anxiety disorders (e.g., separation, social, generalized anxiety disorders), OCD, depression, and substance abuse problems. Exposure therapy is the standard treatment for specific phobia, but many still struggle with symptoms even after treatment. For exposure therapy to be effective, youth with specific phobia must actively approach feared situations to learn that feared outcomes do not occur. Therefore, strategies to facilitate approach behaviors during exposure therapy may improve treatment outcomes.

Self-distancing (SD) is a technique that may help youths approach their fears in exposure therapy. SD utilizes second or third-person language to enhance a person's psychological distance from self, helping them to "take a step back" from emotional situations and adopt a more objective perspective. In community samples, SD has been found to boost determination and persistence during difficult tasks, including those that induce anxiety (e.g., giving a speech). However, SD has yet to be tested as a strategy for helping clinically anxious youth engage with exposures. Additionally, objective measures of approach are needed for measuring and modifying novel exposure therapy augmentation strategies, such as SD, to improve treatment outcomes.

This study will examine if SD increases the ability to approach feared stimuli during a behavioral approach test (BAT). 20 youth (7-12.99 years) with specific phobia of spiders will be randomized to either a SD or a control condition. In the SD condition, participants will engage with the exposure task (BAT) from a self-distanced view (e.g., "Emily will touch a spider"), while in the control condition the subject will use first-person perspective (e.g., "I will touch a spider") Before and after the exposure therapy session, a BAT will be applied. This study will assess: 1) Approach -indexed using both behavioral (ability to get physically closer to spider, and video-derived motion analysis) and neuro-physiological (i.e., electroencephalogram [EEG], heart rate [HR], heart rate variability [HRV] and electrodermal activity [EDA]) metrics, collected during a BAT and 2) severity of specific phobia using validated self-report scales. During SD or control intervention, continuous audio and video data will be collected to derive behavioral metrics of engagement with the intervention (i.e., video-derived motion analysis and audio-derived linguistic metrics) and participants will be asked to subjectively rate their distress and engagement with the activity. Data will be analyzed to determine whether SD improves behavioral, neural, and physiological markers of approach to feared stimuli in youth with specific phobia and reduces symptom severity, and to explore the degree to which changes in video and audio-derived objective metrics of behavioral engagement with the intervention associate with changes in subjective ratings of fear/distress, subjective self-report of engagement and symptom severity.

ELIGIBILITY:
Inclusion Criteria

* Age 7-12.99 years at the time of consent
* Written informed consent by a parent/legal guardian and assent by the child
* Clinically significant symptoms of specific phobia (i.e., spider phobia)
* Fluent in English (Participant may be bilingual but must be able to speak and understand fluent English to participate in the study)

Exclusion Criteria

* Prior diagnosis of bipolar disorder
* Prior diagnosis of psychotic disorders
* Prior diagnosis of autism spectrum disorder
* Active alcohol or substance dependence
* Active suicidal ideation or suicidal behavior within the past 3 months prior to baseline assessment
* Any major medical or neurological problem (e.g., unstable hypertension, seizure disorder, head trauma)
* Any history of cognitive impairment or developmental delay

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Behavioral Approach Test (BAT) | Immediately before and after intervention.
  The BAT will be utilized to evaluate participants' behavioral approach towards a spider before and after the exposure therapy session. Participants will be instructed to approach a spider, contained in a plastic container at the opposite end of the room, as quickly and closely as they can manage, stopping when their fear becomes overwhelming. The BAT outcomes will be assessed by the distance approached (marked on the floor), ranging from 0, where participants will refuse to enter the room or to move from the starting point- to 10 feet, where they will touch the spider with a fingertip.
Spider Phobia Questionnaire (SPQ-C) | At baseline (~1 week before the intervention) and immediately after the intervention.
  The SPQ-C is a validated self-report assessment of spider fear for children 8-12 years, consisting of 29 true/false items, 8 of which are reversed-scored. Total scores range from 0 to 29. Higher scores indicate a greater degree of spider fear.
Treatment Engagement and Adherence Ratings (TEARS) | Immediately after the intervention.
  The TEARS is a brief questionnaire assessing youth and therapist reports of youth's adherence to their assigned exposure condition, and their approach toward the exposure. Adherence and engagement are rated on a Likert scale from 1-7, with higher scores indicating greater engagement and adherence.
Subjective Units of Distress Scale (SUDS) | Immediately before and after the intervention.
  Subjective Units of Distress (SUDs) scale-a self-assessment tool that quantifies the intensity of an individual's distress. During BAT, participants will be asked to indicate their level of anxiety on a scale ranging from 0 "no distress" to 100 "extreme distress".

SECONDARY OUTCOMES:
Heart Rate Variability | Immediately before and after the intervention.
  HRV is a widely recognized indicator of the autonomic nervous system's regulation of the heart, reflecting the body's capacity to adapt to stress and relaxation. HRV has been extensively used in clinical and physiological research to assess cardiovascular function and autonomic engagement.
Electrodermal activity | Immediately before and after the intervention.
  Electrodermal activity (EDA) refers to the changes in the skin's ability to conduct electricity, which is influenced by the activity of the sweat glands. These changes are primarily driven by the sympathetic nervous system, which is activated in response to emotional and physiological arousal. Meta-analyses research suggest that anxious and non-anxious individuals differ in their EDA-estimated fear conditioned responses.
Electroencephalogram (EEG) | Immediately before and after the intervention.
  EEG has become a valuable tool for understanding the neural mechanisms underlying anxiety and phobia, offering high temporal resolution to capture rapid neural responses to fear-related stimuli. Research indicates that increased beta and gamma band activity during exposure to feared stimuli is associated with heightened arousal and fear responses in individuals with specific phobias, while reductions in alpha power are linked to increased anxiety. This outcome will measure the changes in these frequency bands before and after the intervention and compare them with the control condition.

OTHER OUTCOMES:
Screen for Child Anxiety Related Disorders (SCARED)- Parent and Child | At baseline (~1 week before intervention) and immediately after intervention.
  The SCARED is a 41-item measure with parallel forms for youth and caregivers, assessing five domains of anxiety: panic disorder, generalized anxiety disorder, separation anxiety disorder, social anxiety disorder, and school avoidance. It is a well-validated tool with strong psychometric support. Items are rated on a 3-point scale (0 = Not true or hardly ever true, 1 = Somewhat true or sometimes true, 2 = Very true or often true), with total scores ranging from 0 to 82, where higher scores indicate greater anxiety severity.
Child Behavior Checklist (CBCL) | This measure is completed by the child's caregiver at baseline (~1 week before the intervention).
  The Child Behavior Checklist (CBCL) is a widely used parent-report measure that assesses emotional and behavioral problems in children and adolescents (ages 6-18). It consists of 113 items, rated on a 3-point scale (0 = not true, 1 = somewhat true, 2 = very true), with total scores ranging from 0 to 226. Scores are standardized into T-scores, with higher scores indicating greater symptom severity.
Clinical Expectancy Questionnaire (CEQ) | It will be applied immediately before the intervention.
  The Credibility/Expectancy Questionnaire (CEQ) is a validated scale for measuring treatment expectancy and rationale credibility for use in clinical outcome studies. It consists of six items, with credibility items scored from 1 to 9 (range: 3-27) and expectancy items scored from 0% to 100% (range: 0-300%). Scores are typically standardized and analyzed separately for each factor.

CONTACTS AND LOCATIONS:
Overall Officials: Kate D Fitzgerald, MD, Principal Investigator — Professor of Psychiatry
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolitzky-Taylor KB, Horowitz JD, Powers MB, Telch MJ. Psychological approaches in the treatment of specific phobias: a meta-analysis. Clin Psychol Rev. 2008 Jul;28(6):1021-37. doi: 10.1016/j.cpr.2008.02.007. Epub 2008 Mar 7. PMID 18410984
- [Background] Wetzer G, Ten Have M, de Graaf R, Batelaan NM, van Balkom AJLM. Specific Phobia: Risk Factor of Other Psychiatric Disorders. J Nerv Ment Dis. 2021 Jul 1;209(7):484-490. doi: 10.1097/NMD.0000000000001341. PMID 33840768
- [Background] Ollendick, T.H. and N.J. King, Empirically Supported Treatments for Children and Adolescents: Advances Toward Evidence-Based Practice, in Handbook of Interventions that Work with Children and Adolescents. 2004. p. 1-25.
- [Background] Ollendick T, Allen B, Benoit K, Cowart M. The tripartite model of fear in children with specific phobias: assessing concordance and discordance using the behavioral approach test. Behav Res Ther. 2011 Aug;49(8):459-65. doi: 10.1016/j.brat.2011.04.003. Epub 2011 May 6. PMID 21596371
- [Background] Merikangas KR, He JP, Burstein M, Swanson SA, Avenevoli S, Cui L, Benjet C, Georgiades K, Swendsen J. Lifetime prevalence of mental disorders in U.S. adolescents: results from the National Comorbidity Survey Replication--Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry. 2010 Oct;49(10):980-9. doi: 10.1016/j.jaac.2010.05.017. Epub 2010 Jul 31. PMID 20855043
- [Background] Bushnell GA, Gaynes BN, Compton SN, Dusetzina SB, Olfson M, Sturmer T. Incident Substance Use Disorder Following Anxiety Disorder in Privately Insured Youth. J Adolesc Health. 2019 Oct;65(4):536-542. doi: 10.1016/j.jadohealth.2019.05.007. Epub 2019 Jul 17. PMID 31326248
- [Background] Borkovec, T., T. Weerts, and D. Bernstein, Assessment of anxiety in handbook of behavioral assessment. 1997, New York, John Wiley and Sons, Inc.
- [Background] Barzilay R, White LK, Moore TM, Calkins ME, Taylor JH, Patrick A, Huque ZM, Young JF, Ruparel K, Pine DS, Gur RC, Gur RE. Association of anxiety phenotypes with risk of depression and suicidal ideation in community youth. Depress Anxiety. 2020 Sep;37(9):851-861. doi: 10.1002/da.23060. Epub 2020 Jun 5. PMID 32500960
- [Background] Ahlen J, Ghaderi A. Dimension-specific symptom patterns in trajectories of broad anxiety: A longitudinal prospective study in school-aged children. Dev Psychopathol. 2020 Feb;32(1):31-41. doi: 10.1017/S0954579418001384. PMID 30688179